CLINICAL TRIAL: NCT05551832
Title: Prevalence of Marginal Ulcer After PPPD and Preventive Effect of Proton Pump Inhibitor in Korea: A Prospective Multicenter Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Joon Seong Park, professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3-2022-0193
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Pancretic Dissease (Benign/Malignancy); BIle Duct Diseae(Benign/Malignancy); Ampulla of Vater Disease (Benign/Malignancy)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Placebo after Pylurus preserving Pancreaticoduodenctomy (PPPD) for 6 months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo after Pylurus preserving Pancreaticoduodenctomy (PPPD) for 6 months (Placebo Comparator): Placebo beginning day of hospital discharge following PPPD for 6 months
  Interventions: Drug: Arm I (Placebo),
- Esmesol 40mg after PPPD for 6 months (Experimental): Esmesol 40mg beginning day of hospital discharge following PPPD for 6 months
  Interventions: Drug: Arm II (ESMESOL)

INTERVENTIONS:
Drug: Arm I (Placebo), — Placebo after Pylurus preserving Pancreaticoduodenctomy (PPPD) for 6 months
  Arms: Placebo after Pylurus preserving Pancreaticoduodenctomy (PPPD) for 6 months
Drug: Arm II (ESMESOL) — SMESOL 40 mg dose administrea daily at bedtime for 6 months after PPPD ,
  Arms: Esmesol 40mg after PPPD for 6 months

SUMMARY:
This research is to determine which medication, Esmesol (PPI) or Placebo works best at reducing the chance that a patient will get an marginal ulcer after pancreaticoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is age ≥ 19 years Patient meets the criteria for Open/MIS PPPD Females only: Patient is willing to take a urine pregnancy test

Exclusion Criteria:

- Subject allergic to ESMESOL Patient receiving antifungal (i.e. ketoconazole or itraconazole) Hepatic insufficiency History of Crohns disease History of Zollinger-Ellison disease Patient received an investigational drug within 30 days of enrollment Previous Gastric Surgery HX

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Marginal ulcer incidence | Time Frame: during first 6 months after surgery
  Number of Participants occurs Endoscopic visualization of presence or absence of marginal ulcers

SECONDARY OUTCOMES:
QOL | Time Frame: during first 6 months after surgery
  Number of Participants With Complaints, Specifically About Pain, Vomiting, Dyspepsia, and/or Dysphagia.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea